CLINICAL TRIAL: NCT00796757
Title: An Open Label Study of the Effect of First Line Treatment With Avastin (Bevacizumab) in Combination With Low-dose Interferon on Progression-free Survival in Patients With Metastatic Clear Cell Renal Cell Carcinoma.
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Low-Dose-Interferon in Patients With Metastatic Clear Cell Renal Cell Carcinoma (RCC).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO21609; 2007-006611-23
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Interferon alpha-2

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: interferon alfa-2a

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 10mg/kg iv infusion every 2 weeks
Drug: interferon alfa-2a — 3 MIU sc t.i.w.

SUMMARY:
This single arm study will assess progression free survival, tumor response and safety of Avastin in combination with interferon alfa-2a (IFN) as first line treatment in patients with metastatic clear cell renal cell carcinoma. Patients will receive Avastin (10mg/kg iv) every 2 weeks in combination with a low dose of interferon alfa-2a (3 MIU sc three times per week (t.i.w.). The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* metastatic RCC with majority (>50%) of conventional clear-cell type;
* prior total nephrectomy for primary RCC;
* at least one measurable or non-measurable lesions;
* ECOG performance score of 0 or 2.

Exclusion Criteria:

* prior systemic treatment for metastatic RCC;
* current or previously treated but non-stable CNS metastases or spinal cord compression;
* major surgery (including open biopsy) or radiation therapy within 28 days prior to enrollment;
* significant cardiovascular disease within 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2008-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- Czechia (2):
  - Olomouc
  - Prague
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (2):
  - Seinäjoki
  - Turku
- Germany (12):
  - Arnsberg
  - Augsburg
  - Berlin
  - Freiburg im Breisgau
  - Homburg/Saar
  - Leipzig
  - München
  - Münster
  - Offenburg
  - Planegg
  - Stuttgart
  - Weiden
- Greece (2):
  - Larissa
  - Thessaloniki
- Italy (3):
  - Milan
  - Napoli
  - Pisa
- Lithuania (2):
  - Kaunas
  - Vilnius
- Netherlands (4):
  - Amstelveen
  - Eindhoven
  - Maastricht
  - Nijmegen
- Russia (7):
  - Barnaul
  - Moscow
  - Obninsk
  - Saint Petersburg
  - Ufa
  - Ulyanovsk
  - Yekaterinburg
- Sweden (4):
  - Eskilstuna
  - Linköping
  - Sundsvall
  - Vaxjo
- Switzerland (3):
  - Aarau
  - Locarno
  - Zurich
- United Kingdom (2):
  - Cambridge
  - Cardiff

REFERENCES:
- [Derived] Melichar B, Bracarda S, Matveev V, Alekseev B, Ivanov S, Zyryanov A, Janciauskiene R, Fernebro E, Mulders P, Osborne S, Jethwa S, Mickisch G, Gore M, van Moorselaar RJ, Staehler M, Magne N, Bellmunt J; BEVLiN Investigators. A multinational phase II trial of bevacizumab with low-dose interferon-alpha2a as first-line treatment of metastatic renal cell carcinoma: BEVLiN. Ann Oncol. 2013 Sep;24(9):2396-402. doi: 10.1093/annonc/mdt228. Epub 2013 Jun 26. PMID 23803225

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab Plus (+) Interferon: Participants received bevacizumab 5 milligrams per kilogram (mg/kg) intravenously (IV) on Day 1 and Interferon alpha-2a (IFN) 3 million international units (MIU) subcutaneously (SC) 3 times per week with at least 1 day between injections. This cycle lasted for 2 weeks and was repeated until disease progression, unacceptable toxicity, or participant withdrawal.
Period: Overall Study
Arm/Group | Bevacizumab Plus (+) Interferon
Started | 146
Completed | 60
Not Completed | 86
Not completed — Withdrawal by Subject | 14
Not completed — Death | 61
Not completed — Protocol Violation | 1
Not completed — Participant noncompliance | 1
Not completed — Investigator's decision | 2
Not completed — Other | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of either or both study drugs and had a valid baseline assessment and at least 1 postbaseline assessment.
Groups:
- Bevacizumab + Interferon: Participants received bevacizumab 5 mg/kg IV on Day 1 and IFN 3 MIU SC 3 times per week with at least 1 day between injections. This cycle lasted for 2 weeks and was repeated until disease progression, unacceptable toxicity, or participant withdrawal.
Arm/Group | Bevacizumab + Interferon
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 98

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) - Percentage of Participants Estimated to be Progression Free at 12 and 24 Months
Description: PFS at 12 and 24 months is an estimate of the percentages of participants expected to be progression free at 12 and 24 months based on Kaplan-Meier survival analysis of the PFS data. PFS was defined as the time period from the first postbaseline tumor assessment to evidence of disease progression or death from any cause, whichever occurred first. Disease progression included evaluation solely due to symptomatic deterioration or death due to any reason. Censoring at start of any subsequent antineoplastic therapy was not performed.
Time Frame: 12 and 24 months
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Interferon
Number analyzed (Participants) | 146
percentage of participants
  12 months | 58.2 [49.9 to 66.6]
  24 months | 28.9 [20.8 to 36.9]

2. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Reponse (CR) or Partial Response (PR)
Description: Percentage of participants with objective response, termed responders, based assessment of confirmed CR or confirmed PR according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses were those that persisted on repeat imaging study greater than or equal to (≥)4 weeks after initial documentation of response. CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must have decreased to normal (short axis less than [<]10 millimeters [mm]). No new lesions. PR was defined as ≥30 percent (%) decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Baseline, every 8 weeks to Week 32 then every 12 weeks to disease progression or a maximum of 2 years from enrollment of last participant
Population: ITT population; only participants with measurable disease were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Interferon
Number analyzed (Participants) | 139
percentage of participants | 28.8

3. Primary Outcome: PFS - Percentage of Participants With an Event
Description: PFS was defined as the time period from the first postbaseline assessment tumor assessment to evidence of disease progression or death from any cause, whichever occurred first. Disease progression included evaluation solely due to symptomatic deterioration or death due to any reason. Censoring at start of any subsequent antineoplastic therapy was not performed.
Time Frame: as for outcome 2
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Interferon
Number analyzed (Participants) | 146
percentage of participants | 69.2

4. Primary Outcome: PFS - Time to Event
Description: as for outcome 3
Time Frame: as for outcome 2
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Interferon
Number analyzed (Participants) | 146
months | 15.3 [11.7 to 18.0]

5. Secondary Outcome: Overall Survival (OS) - Percentage of Participants Estimated to be Alive at 12 and 24 Months
Description: OS at 12 and 24 months is the estimate of the percentages of participants expected to alive at 12 and 24 months based on Kaplan-Meier survival analysis of the survival data. Median OS was defined as the time period from the first bevacizumab infusion to death from any cause. Censoring at start of any subsequent antineoplastic therapy was not performed.
Time Frame: Day 0, every 2 weeks until disease progression or end of treatment visit (28 days after last bevacizumab infusion, every 3 months during follow-up, or a maximum of 2 years from enrollment of last participant
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Interferon
Number analyzed (Participants) | 146
percentage of participants
  12 months | 84.1 [78.0 to 90.2]
  24 months | 59.6 [51.0 to 68.2]

6. Secondary Outcome: OS - Percentage of Participants With an Event
Description: OS was defined as the time period from the first bevacizumab infusion to death from any cause. Censoring at start of any subsequent antineoplastic therapy was not performed.
Time Frame: as for outcome 5
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Interferon
Number analyzed (Participants) | 146
percentage of participants | 41.8

7. Secondary Outcome: OS - Time to Event
Description: as for outcome 6
Time Frame: as for outcome 5
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Interferon
Number analyzed (Participants) | 146
months | 30.7 [25.7 to NA] — The upper limit of the 95% confidence interval (CI) could not be estimated because the follow-up time was too short to observe enough survival events for complete data estimation.

8. Secondary Outcome: Percentage of Participants With Any Health Problems as Assessed by the European Quality of Life 5 Dimensions (EQ-5D) by Visit
Description: EQ-5D is a standardized, participant-administered measure of health outcome. It provides a descriptive profile for 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), using 3 levels (no, moderate, or extreme problems) and a single index value characterizing current health status using a 100-point visual analog scale (0=worst, 100=best). Answers from the questionnaire for each dimension (mobility, self-care, usual activity, pain/discomfort, and anxiety/depression) was classified into one of 2 categories: 'no problems' or 'any problems', and the percentage of participants in each category was determined.
Time Frame: Screening/Baseline, Cycle 7, Cycle 25, Cycle 43, Cycle 61, and End of Treatment (EOT)
Population: ITT population; number (n) equals (=) number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Interferon
Number analyzed (Participants) | 145
percentage of participants
  Mobility, no problems, Baseline (n=142) | 69.0
  Mobility, any problems, Baseline (n=142) | 31.0
  Mobility, no problems, Cycle 7 (n=106) | 64.2
  Mobility, any problems, Cycle 7 (n=106) | 35.8
  Mobility, no problems, Cycle 25 (n=69) | 58.0
  Mobility, any problems, Cycle 25 (n=69) | 42.0
  Mobility, no problems, Cycle 43 (n=36) | 38.9
  Mobility, any problems, Cycle 43 (n=36) | 61.1
  Mobility, no problems, Cycle 61 (n=22) | 40.9
  Mobility, any problems, Cycle 61 (n=22) | 59.1
  Mobility, no problems, EOT (n=82) | 41.3
  Mobility, any problems, EOT (n=82) | 58.8
  Self-care, no problems, Baseline (n=145) | 82.8
  Self-care, any problems, Baseline (n=145) | 17.2
  Self-care, no problems, Cycle 7 (n=106) | 81.1
  Self-care, any problems, Cycle 7 (n=106) | 18.9
  Self-care, no problems, Cycle 25 (n=69) | 81.2
  Self-care, any problems, Cycle 25 (n=69) | 18.8
  Self-care, no problems, Cycle 43 (n=36) | 69.4
  Self-care, any problems, Cycle 43 (n=36) | 30.6
  Self-care, no problems, Cycle 61 (n=22) | 77.3
  Self-care, any problems, Cycle 61 (n=22) | 22.7
  Self-care, no problems, EOT (n=80) | 63.8
  Self-care, any problems, EOT (n=80) | 36.3
  Usual activity, no problems, Baseline (n=145) | 60.7
  Usual activity, any problems, Baseline (n=145) | 39.3
  Usual activity, no problems, Cycle 7 (n=106) | 53.8
  Usual activity, any problems, Cycle 7 (n=106) | 46.2
  Usual activity, no problems, Cycle 25 (n=69) | 46.4
  Usual activity, any problems, Cycle 25 (n=69) | 53.6
  Usual activity, no problems, Cycle 43 (n=36) | 33.3
  Usual activity, any problems, Cycle 43 (n=36) | 66.7
  Usual activity, no problems, Cycle 61 (n=22) | 45.5
  Usual activity, any problems, Cycle 61 (n=22) | 54.5
  Usual activity, no problems, EOT (n=78) | 33.3
  Usual activity, any problems, EOT (n=78) | 66.7
  Pain/discomfort, no problems, Baseline (n=145) | 48.3
  Pain/discomfort, any problems, Baseline (n=145) | 51.7
  Pain/discomfort, no problems, Cycle 7 (n=106) | 49.1
  Pain/discomfort, any problems, Cycle 7 (n=106) | 50.9
  Pain/discomfort, no problems, Cycle 25 (n=69) | 53.6
  Pain/discomfort, any problems, Cycle 25 (n=69) | 46.4
  Pain/discomfort, no problems, Cycle 43 (n=36) | 50.0
  Pain/discomfort, any problems, Cycle 43 (n=36) | 50.0
  Pain/discomfort, no problems, Cycle 61 (n=22) | 50.0
  Pain/discomfort, any problems, Cycle 61 (n=22) | 50.0
  Pain/discomfort, no problems, EOT (n=80) | 33.8
  Pain/discomfort, any problems, EOT (n=80) | 66.3
  Anxiety/depression, no problems, Baseline (n=144) | 45.8
  Anxiety/depression, any problems, Baseline (n=144) | 54.2
  Anxiety/depression, no problems, Cycle 7 (n=106) | 55.7
  Anxiety/depression, any problems, Cycle 7 (n=106) | 44.3
  Anxiety/depression, no problems, Cycle 25 (n=69) | 62.3
  Anxiety/depression, any problems, Cycle 25 (n=69) | 37.7
  Anxiety/depression, no problems, Cycle 43 (n=36) | 61.1
  Anxiety/depression, any problems, Cycle 43 (n=36) | 38.9
  Anxiety/depression, no problems, Cycle 61 (n=22) | 59.1
  Anxiety/depression, any problems, Cycle 61 (n=22) | 40.9
  Anxiety/depression, no problems, EOT (n=80) | 45.0
  Anxiety/depression, any problems, EOT (n=80) | 55.0

9. Secondary Outcome: EQ-5D - Visual Analog Scale (VAS)
Description: EQ-5D: participant-rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 millimeters (mm) (best imaginable health state); higher scores indicate a better health state. Participants were asked to rate their health state and mark the line; the distance from the left edge was recorded. For change from baseline a negative value represents a worsening in the health state and a positive value represents an improvement in the health state.
Time Frame: Screening/Baseline, Cycle 7, Cycle 25, Cycle 43, Cycle 61, and EOT
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bevacizumab + Interferon
Number analyzed (Participants) | 140
mm
  Baseline (n=140) | 71.2 (17.27)
  Cycle 7 (n=103) | 71.8 (13.63)
  Change at Cycle 7 (n=99) | -1.8 (14.54)
  Cycle 25 (n=68) | 72.4 (15.46)
  Change at Cycle 25 (n=67) | -2.3 (17.84)
  Cycle 43 (n=36) | 71.3 (17.12)
  Change at Cycle 43 (n=36) | -0.9 (20.12)
  Cycle 61 (n=22) | 70.5 (15.74)
  Change at Cycle 61 (n=22) | -1.7 (20.41)
  EOT (n=79) | 65.2 (19.72)
  Change at EOT (n=77) | -7.7 (15.73)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the date of first administration of bevacizumab until 28 days after the last administration of bevacizumab and/or IFN.
Description: All Grade >3 AEs documented. Only Grade 1/2 AEs related to bevacizumab and/or IFN occurring from first bevacizumab administration up to 28 days after last dose were documented.
Arm/Group | Bevacizumab + Interferon
Serious Adverse Events (participants affected / at risk) | 26/146
Other Adverse Events (participants affected / at risk) | 113/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Interferon (N=146)
Abscess (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular stenosis (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Asthenia (General disorders) | 3
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Depression (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Hypertension (Vascular disorders) | 2
Overdose (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Interferon (N=146)
Pyrexia (General disorders) | 28
Fatigue (General disorders) | 41
Asthenia (General disorders) | 15
Chills (General disorders) | 13
Nausea (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 10
Stomatitis (Gastrointestinal disorders) | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20
Hypertension (Vascular disorders) | 51
Decreased appetite (Metabolism and nutrition disorders) | 17
Headache (Nervous system disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Neutropenia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 10
Nasopharyngitis (Infections and infestations) | 8
Proteinuria (Renal and urinary disorders) | 63
Weight decreased (Investigations) | 8
Blood creatinine increased (Investigations) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request the Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.